CLINICAL TRIAL: NCT00605670
Title: Measuring Patient Satisfaction and Quality of Life Following Body Image Altering Surgery: Development and Validation of a Patient-Reported Outcomes Instrument
Brief Title: Measuring Patient Satisfaction and Quality of Life Following Body Image Altering Surgery
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: McMaster University (Other); University College, London (Other); Dartmouth-Hitchcock Medical Center (Other); University of British Columbia (Other); Johns Hopkins University (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 05-058
Record Dates: First submitted 2008-01-11; First posted 2008-01-31 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer; Breast Surgery; Breast Reconstruction; Breast Reduction; Breast Augmentation
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Postoperative Breast Surgery Patients
  Interventions: Behavioral: questionnaires
- 2: Preoperative Breast Surgery Patients
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — patients will fill out two questionnaires post surgery
  Groups: 1
Behavioral: questionnaires — Patient will fill out questionnaire before and 3 to 6 months after treatment.
  Groups: 2

SUMMARY:
The goal of this study is to develop a questionnaire to measure patient satisfaction with their breast surgery. This questionnaire will help surgeons better understand how patients feel about their surgical results. We hope that such a questionnaire will improve the understanding of breast surgery results and patient care.

ELIGIBILITY:
Inclusion Criteria:

* All stages (1-4)
* Age > or = to 18 to 85 years.
* Postoperative Group: Male and Female patients who have undergone mastectomy, breast reconstruction, reduction, augmentation, bariatric or body contouring surgery between 1 month to 8 years ago

Or

* Preoperative Group: Male and Female patients who are scheduled to undergo mastectomy, breast reconstruction, reduction, or augmentation or body contouring surgery

Exclusion Criteria:

* Inability to speak or understand English
* Active psychiatric illness, cognitive or sensory impairment
* Physical impairment that may prevent filling out a paper and pencil survey or responding to interview questions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinics at the various sites
Sampling Method: Non-Probability Sample
Enrollment: 722 (Actual)
Dates: Start 2005-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To develop and validate a new patient derived measure of satisfaction with breast surgery. | conclusion of study

SECONDARY OUTCOMES:
Determining variations in satisfaction related to patient characteristics and preoperative expectations. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pusic, M.D., M.H.S., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (4):
  - John Hopkins Medical Center, Baltimore, Maryland
  - Dartmouth Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org